CLINICAL TRIAL: NCT03562585
Title: Immunological Measurement of Aspartate/Alanine Aminotransferase Utilizing Monoclonal Anti-bodies in Predicting Liver Fibrosis and Inflammation
Brief Title: Immunological Measurement of Aspartate/Alanine Aminotransferase
Status: Completed | Type: Observational
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Ki Tae Suk, Hallym university College of Medicine, Chuncheon Sacred Heart Hospital
Other Study IDs: ASTALT
Record Dates: First submitted 2018-05-13; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Chronic Liver Disease and Cirrhosis
Keywords: Chronic hepatitis B; Alanine Aminotransferase; Aspartate Aminotransferase
MeSH Terms: conditions — Fibrosis; Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Efficacy of immunoassay in liver fibrosis: efficacy of immunoassay in liver fibrosis in patients with CHB
  Interventions: Diagnostic Test: with sandwich ELISA immunoassay with fluorescence labeled monoclonal antibodies

INTERVENTIONS:
Diagnostic Test: with sandwich ELISA immunoassay with fluorescence labeled monoclonal antibodies — with sandwich ELISA immunoassay with fluorescence labeled monoclonal antibodies

SUMMARY:
Previous reports have suggested that ALT-immunoglobulin complex was increased according to the severity of the liver disease, and high concentration of mAST and this might indicate a severely damaged liver. Immunoassay might be useful as a screening method in the differ-ential diagnosis of liver fibrosis according to patients. In this study, the efficacy of immunoas-say in the prediction of liver fibrosis in patients with chronic hepatitis B (CHB) was evaluated.

DETAILED DESCRIPTION:
Enzymatic analysis of aspartate/alanine aminotransferase (AST/ALT) does not exactly represent the progression of liver fibrosis. Immunoassay for the AST (cytoplasmic [c] AST/mitochondrial [m] AST) and ALT (ALT1/ALT2) have been suggested as one of the alternatives for the enzy-matic analysis. We evaluated the efficacy of immunoassay in predicting liver fibrosis and in-flammation. A total of 219 patients with chronic hepatitis B (CHB) who underwent hepatic ve-nous pressure gradient (HVPG) and liver biopsy before antiviral therapy were recruited. Serum samples were prepared from blood during HVPG. The liver function test including enzymatic AST/ALT and immunological cAST, mAST, ALT1 and ALT2 were checked with sandwich ELI-SA immunoassay with fluorescence labeled monoclonal antibodies, and were compared with the METAVIR stage of live fibrosis and the Knodell grade of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* patients with CHB, who simultaneously underwent HVPG and liver biopsy for the routine check-up prior to antiviral treatment, were prospectively recruited.

Exclusion Criteria:

* Patients were selected according to inclusion criteria with CHB and then excluded according to exclusion criteria: i. they had other cause with liver disease: ii. decompensated cirrhosis and re-ceived antiviral treatment within the previous 6 months. iii. malignancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between January 2007 and December 2010, patients with CHB, who simultaneously underwent HVPG and liver biopsy for the routine check-up prior to antiviral treatment, were prospectively recruited.
  They are all admitted for the evaluation of CHB. Age: 20-70 Gender: both, Korean
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2010-12-30 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
A sandwich enzyme immune-assay (ALT1, ALT2, mAST, cAST) according to fibrosis and inflammation | 3 years
  efficacy of immunoassay in predicting liver fibrosis and inflammation.

SECONDARY OUTCOMES:
HVPG score | 3 years
  efficacy of HVPG in predicting liver fibrosis and inflammation.